CLINICAL TRIAL: NCT03865563
Title: Selective Transvenous Chemoembolization of Primary Pancreatic Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We need to make significant adjustments to proposed drug and its delivery method
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1936; IRB00164996 (Other: JHM IRB)
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: retrograde venous infusion; chemotherapy; gemcitabine; lipiodol
MeSH Terms: interventions — Ethiodized Oil

STUDY DESIGN:
Intervention Model Description: This is an open-label, single institution, single-arm pilot study, designed to assess the feasibility, safety and efficacy of retrograde venous infusion of gemcitabine/Lipiodol® administered in a neoadjuvant setting for the treatment of patients with resectable, borderline-resectable or locally-advanced pancreatic adenocarcinoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pancreatic adenocarcinoma (Experimental): Participants with resectable, borderline-resectable or locally-advanced pancreatic adenocarcinoma will receive pancreatic retrograde venous infusion of gemcitabine/lipiodol
  Interventions: Drug: Retrograde venous infusion of gemcitabine/lipiodol

INTERVENTIONS:
Drug: Retrograde venous infusion of gemcitabine/lipiodol — Access will be gained into the portal vein via a transhepatic approach. The pancreatic tumor-draining veins will be accessed via a catheter positioned in the portal vein, superior mesenteric vein or splenic vein. The catheter is then advanced into the vein draining the segment in which the targeted tumor is located. Tumor location and its venous drainage will be confirmed with sub-selective pancreatic venography and cone-beam CT. Once correct catheter positioning is confirmed, the gemcitabine/Lipiodol® emulsion will be administered under real-time fluoroscopic guidance until the entire dose is administered or until stasis is achieved in the vein through which the drug is being delivered.
  Other Names: Pancreatic retrograde venous infusion (PRVI)

SUMMARY:
Catheter directed retrograde venous infusion of gemcitabine/lipiodol into pancreatic tumors.

DETAILED DESCRIPTION:
Overall, subjects with resectable, borderline-resectable and/or locally-advanced pancreatic cancer are eligible to be entered into the study. Each enrolled study subject will receive a single neoadjuvant pancreatic retrograde venous infusion (PRVI) administration of the gemcitabine/Lipiodol® emulsion.

Complete enrollment in 12 months from date of enrollment of first study subject.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pathologically and radiologically-confirmed pancreatic adenocarcinoma confined to the pancreas with initial diagnosis within 8 weeks of consent
* Resectable, borderline-resectable or locally-advanced primary pancreatic adenocarcinoma per NCCN guidelines
* The patient is deemed a candidate for the study by the Johns Hopkins Multidisciplinary Pancreatic Tumor Board
* Preserved liver function (Child-Pugh A-B class) without significant liver decompensation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at study entry
* Measurable or evaluable disease that will be directly treated with intra-pancreatic therapy (as defined by Response Evaluation Criteria in Solid Tumors [RECIST 1.1]
* Suitable for PRVI, based on blood parameters such as platelet count, LFTs including bilirubin and coagulation status including international normalized ratio (see "Exclusion Criteria" below)
* The patient is able to give informed consent
* The patient, if a woman of childbearing potential, has a negative pregnancy test
* The patient is willing and able to comply with study procedures, scheduled visits, and treatment plans
* Life expectancy of at least 3 months

Exclusion Criteria:

* Serum total bilirubin > 3.0 mg/dL
* Creatinine > 2.0 mg/dL
* Platelets < 75,000/μL
* Hgb < 8.0 g/dl
* ANC ≤ 1,000/μL
* INR > 2.0
* Complete portal vein thrombosis or significant cavernous transformation of the portal vein
* Ascites (trace ascites on imaging is OK)
* The patient is pregnant or breast-feeding
* The patient is allergic to contrast media that cannot be readily managed or prevented with premedication
* Patients with peripheral neuropathy [> grade 1, according to the National Cancer Institute Common Toxicity Criteria v5.0 (CTAE v5.0)]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility as determined by technical success of Pancreatic Retrograde Venous Infusion (PRVI) with gemcitabine and Lipiodol® | 30 days
  Technical success is measured as number of participants who did not experience technical failure, which is defined as the inability to administer the gemcitabine/ Lipiodol® to the targeted pancreatic tumor.
Safety as measured by number of participants with Grade 3, 4, and 5 toxicities | 30 days
  Number of participants with Grade 3, 4, and 5 toxicities as defined by the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; Version 5.0) that occur during and within 30 days after PRVI

SECONDARY OUTCOMES:
Efficacy as assessed by Objective tumor response | 30 days
  Objective tumor response is measured as number of participants with response as determined by RECIST 1.1 criteria to assess change in tumor size and percent tumor enhancement as visualized on pancreatic protocol CT scans.
Efficacy as assessed by change in serum CA19-9 | Change from baseline to 30 days
  Change in serum CA19-9 measurements pre- and post-PRVI.
Efficacy as assessed by change in levels of gemcitabine and dFdu in peripheral blood samples | Change from baseline to 30 days
  Change in levels of gemcitabine and its inactive metabolite 2',2'-Difluorodeoxyuridine (dFdU) found in peripheral blood samples pre-and post-PRVI.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Liddell, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No